CLINICAL TRIAL: NCT04471961
Title: Analyse of Tumour and Constitutional DNA for the Study of the Determinism in Child Neoplasia
Acronym: ALADIN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Soroptimist association of Monaco (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RECHMPL19_0519; 2020-A0298-31 (Other: IDRCB)
Record Dates: First submitted 2020-07-10; First posted 2020-07-15 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Pediatric Tumor; Familial Cancer; Solid Tumor, Childhood; Hematological Tumor
Keywords: Pediatric oncology; Exome based trio; Cancer predisposition gene; Target therapies; Tumor exome; Transcriptome
MeSH Terms: conditions — Neoplasms; Hematologic Neoplasms | interventions — Exome Sequencing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Children with cancer (Proband) with theirs parents (Experimental)
  Interventions: Genetic: Exome sequencing in pediatrics cancers

INTERVENTIONS:
Genetic: Exome sequencing in pediatrics cancers — This pediatric oncology study proposing a global approach integrating trio-based whole exome sequencing, somatic DNA and RNA analysis will improve the recognition of genetic predisposition and the characterization of target therapies in children with cancer.

SUMMARY:
Background. Cancer is the leading cause of death by disease in children. Most pediatric tumors differ from adult tumors in terms of biological and clinical characteristics. In children, the part of genetic determinism could be higher since the role of environmental factors may be less pronounced than in adults and that a young age at onset is a main feature of genetic cancer predisposition. Recent studies suggested that a number of genetic predisposition remains to be characterized.

Methods. Trio-Based whole exome sequencing of germline DNA from patients (children and adults diagnosed with cancers between 0 and 17 years) and parents will be performed prospectively in a multicentric study including 40 unselected cases of malignant tumor. Participating hospitals will include the CHU of Montpellier, the CHU de Nice and the AP-HP. Tumor analysis will include whole exome analysis and transcriptome for the identification of therapeutic target and contribute to confirm potential link between constitutive mutations and tumor phenotype (such as loss of expression, loss of heterozygosity).

Perspectives. This pediatric oncology study proposing a global approach integrating trio-based whole exome sequencing, somatic DNA and RNA analysis will improve the recognition of genetic predisposition and the characterization of target therapies in children with cancer.

ELIGIBILITY:
Inclusion Criteria:

* The patient has a solid or haematological malignancy, either familial forms or isolated cases diagnosed between the ages of 0 and 17 years.
* The minor patient and both biological parents are available to participate in the study OR
* The adult patient and one or both parents are available to participate in the study.
* The patient's parents must have given their free and informed consent and signed the consent for the minor's participation in the study.
* The patient's parent(s) must have given free and informed consent and the patient of legal age must have signed the consent for participation in the study.
* The patient must be affiliated or beneficiary of a Frrench social security scheme.

Exclusion Criteria:

* The patient's parents are under guardianship or trusteeship or under legal protection Yes No
* Failure to obtain written informed consent from parents (for themselves and their minor child) after a period of reflection Yes No
* No affiliation to or beneficiary of a French social security scheme (for biological parents and the patient)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-07-09 (Actual); Primary Completion 2025-02-12 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification of genetic variants and confirmation of the causality of these variants for the patient's pathology whole exome sequencing | 12 months
  A blood sample will be taken from patients and their parents in order to carry out genetic analyses.
  New generation NGS Exome sequencing in trio (patient and 2 healthy parents) on an Illumina HiSeq 2000 platform using the SureSelectXT Human All Exon 50Mb, V5 kit.
  Bioinformatics analysis of the data. Confirmation of mutations by Sanger sequencing (gold standard).
  In case of identification of mutations in candidate genes confirmed by Sanger sequencing, we will perform functional and clinical-genetic studies.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Pujol, PU-PH, Principal Investigator — Montpellier University Hospital
Locations (1):
- CHU Montpellier, Montpellier, Occitanie, France